CLINICAL TRIAL: NCT06268470
Title: Efficacy of Antiplatelet Therapy for the Treatment of Chronic Recalcitrant Urticaria
Brief Title: Antiplatelet Therapy in Chronic Urticaria
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Jettanong Klaewsongkram, MD., Assoc. Prof. Jettanong Klaewsongkram, MD., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chula-ARC 001/18
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria; antiplatelet; D-dimer
MeSH Terms: conditions — Chronic Urticaria | interventions — desloratadine; Cilostazol; Dipyridamole; Histamine Antagonists

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with chronic urticaria will be assigned to 2 treatment arms. 1. high dose antihistamine with antiplatelets; and 2. high dose antihistamine alone.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Identical capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desloratadine (Active Comparator): Oral desloratadine 20 mg/day (antihistamine) for 4 weeks
  Interventions: Drug: Desloratadine
- Desloratadine plus cilostazol and dipyridamole (Experimental): Oral desloratadine 20 mg/day (antihistamine) in conjunction with cilostazol 150 mg/day and dipyridamole 50 mg/day (antiplatelets) for 4 weeks
  Interventions: Drug: Desloratadine plus cilostazol and dipyridamole; Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine plus cilostazol and dipyridamole — Desloratadine 20 mg/day plus cilostazol 150 mg/day and dipyridamole 50 mg/day
  Other Names: Antihistamine plus antiplatelets
  Arms: Desloratadine plus cilostazol and dipyridamole
Drug: Desloratadine — Desloratadine 20 mg/day
  Other Names: Antihistamine alone

SUMMARY:
This study compares the combination of antiplatelets and antihistamine versus antihistamine alone for the treatment of chronic spontaneous urticaria

DETAILED DESCRIPTION:
This study is a randomized control trial comparing the effectiveness of the combination of antiplatelets and antihistamine and antihistamine alone for the treatment of chronic spontaneous urticaria

ELIGIBILITY:
Inclusion Criteria:

Chronic spontaneous urticaria

D-dimer levels over 500 ng/ml

Not respond to a conventional dose of antihistamine

Exclusion Criteria:

Are taking aspirin

Have bleeding tendency

Have concurrent severe medical illnesses

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Weekly urticaria activity score | 4 weeks
  Urticaria activity score over 7 days (UAS7): scores 0-42 from mild to severe

SECONDARY OUTCOMES:
D-dimer levels | 4 weeks
  D-dimer levels

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No